CLINICAL TRIAL: NCT06420141
Title: The Prevalence of Neuropathic Pain Pathophysiology Associated With Ankle Fracture
Acronym: AFNP
Status: Recruiting | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Roman M. Natoli, Associate Professor of Anesthesia, Indiana University
Other Study IDs: 19914
Record Dates: First submitted 2024-03-04; First posted 2024-05-17 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fracture Group: patients with qualifying ankle fractures
- Control Group: Healthy controls without an ankle fracture

SUMMARY:
This application addresses the Peer Reviewed Medical Research Program Investigator-Initiated Research Award FY21 W81XWH-22-CPMRP-IIRA area of Chronic Pain Management Research Program- The investigators will utilize subjects who have sustained ankle fractures and may develop chronic pain following bone union. No attempt will be made to affect the experimental outcome in the subjects. This study will adhere to a core set of standards for rigorous study design and reporting to maximize the reproducibility and translational potential of research.

DETAILED DESCRIPTION:
Persistent pain following bone fracture, such as neuropathic pain (NP), is a possible outcome of fracture repair following injury to the ankle and exhibits incidence rates at 1-year post-surgery of 18-42%. This pain state following bone healing (also known as bone union) will be referred to as bone fracture-associated NP (BFNP). Ankle fractures are among the most common surgically-treated fractures in adults, with the greatest incidence occurring in young males. Women are more commonly affected in other age groups. Distal radius fractures are the most common type of fracture for all age groups. Full healing from a fracture can take anywhere from several weeks to months. Pain that persists after fracture union has taken place is called chronic pain. Chronic or persistent NP is one of the worst, longest-lasting, and difficult symptom to manage after fracture repair in civilian and military populations. It is likely that some of the mechanisms leading to BFNP propagate early after injury, leading to opportunity for early interventions to prevent chronic pain.

NP associated with bone fracture originates from an injury affecting the sensory aspects of the peripheral nervous system and may be associated with abnormal sensations called dysesthesia or from normally non-painful stimuli (allodynia). The condition may have continuous and/or episodic (paroxysmal) components, with the latter resembling stabbing pain or electric shocks. The condition of NP also tends to affect defined dermatomes, and there may be limits to the area of pain. The general working principle is that the injury leading to pain must directly involve the nociceptive pathways. An additional element which can contribute to NP includes sensitization of intact, uninjured pain neurons, which innervate the region adjacent to injured nerve fibers. These changes in the uninjured neurons may induce ongoing pain and may account for certain aspects of hyperalgesia (increased sensitivity to feeling pain). Conditions associated with bone fracture-associated NP (BFNP) include traction neuropathy, nerve compression from soft tissue edema, bone fragment, implants, and/or hematoma.

In civilian adult populations, prevalence rates of NP are about 1 in every 10 adults over age 30, though the prevalence rate and people identified vary depending on the method of identification of NP. Though not distinctly defined as NP due to bone fracture, active-duty personnel and Veterans are at an increased risk of severe pain conditions compared with civilians. Given the numbers of active duty and Veterans who experience pain due to injury, the US military instituted a number of programs, guidelines and initiatives to better manage acute pain for combat-related injuries. These programs include pain control methods which can be readily administered and provide pain relief during immediate field hospital care, transport and subsequent care at military treatment facilities. Despite the instituted practices by the military, BFNP after fracture is a major problem and the literature that documents detailed outcomes of BFNP data are scarce.

Bone fracture is known to induce a complex post-fracture healing process and involves an extensive inflammatory response by immune cells. These immune cells proliferate and permeate the fracture site and secrete a range of pro-inflammatory cytokines which aid in the healing process. However, some of these same proteins are known to contribute to a variety of pain conditions/diseases including migraine, fibromyalgia, complex regional pain syndrome and neuropathic pain. To better understand the manner in which immune cell production of factors contribute to chronic pain states, the investigaotrs have embarked on a series of clinical investigations of immune cells which may contribute to chronic post-traumatic headache following mild traumatic brain injury. Like previous work by other groups, the investigators have observed a unique response by immune cell subsets that may serve to discriminate between both subacute and chronic events following traumatic injury. These attributes may prove to be diagnostic and could be regarded as a hallmark of the development of BFNP by ultimately influencing pain modulation in the clinical patient. Additional mechanisms which may contribute to BFNP include a wind-up of mechanisms in the spinal cord (central sensitization), and maladaptive neuroplasticity with changes in endogenous pain modulation. Anti-nociceptive endogenous pain modulation involves intact engagement of descending pain inhibitory pathways, which serve to protect the injured individual from transforming acute pain to a chronic pain state. However, inefficient descending pain inhibition can be a pathogenic risk factor for developing chronic pain. The degree to which an individual can be assayed for an intact endogenous pain inhibition system can be assessed using a quantitative sensory test (QST) which serves to test condition pain modulation (CPM). The provoking factor for such a generalized sensitization of the pain system could be the continuous noxious input in earlier phases of the bone fracture healing process associated with the ongoing states of inflammation.

Outcomes after trauma which contribute to chronic pain states are complex and are highlighted by a generalized failure in the clinical arena to improve patient conditions and quality of life once these conditions manifest themselves within the individual. However, recent studies have begun to yield novel insights into the injury-associated immune response which may be central to BFNP by using computational methods that account for temporal and spatial networks of mediators. Fundamental understanding of the immunologic responses associated with BFNP at distinct cross-sections in the recovery time frame and dynamically during progression of fracture healing process may yield better management and potentially mitigation of BFNP. Moreover, changing the standard of care treatment for BFNP by identifying at-risk patients early after injury could lead to decreased economic burden in treating BFNP and mitigation of the substantial decrease in quality of life these patients experience. Thus, evidenced-based and "precision" approaches to BFNP and management are greatly needed, in which mechanisms and other factors that contribute to BFNP are identified to guide treatment. The proposed project is significant because it is an essential step in understanding whether ankle fracture chronically alters biological pain risk factors. Such information is critical to 1) developing effective strategies to reduce the occurrence of BFNP, 2) providing prognostic information to individuals suffering with BFNP, and 3) designing evidenced-based and personalized treatments for BFNP.

The proposed study is innovative because it will be the first prospective human study to evaluate the impact of bone fracture on innate immune function and endogenous pain modulatory function across time. This novel information will enhance our understanding of how ankle fracture elicits pathological risk factors for BFNP. Identification of salient risk factors for the initiation and maintenance of BFNP will allow a more personalized injury prognosis to predict those at greatest risk.

ELIGIBILITY:
Fracture Group:

Inclusion Criteria:

1. 18-85 years old
2. an isolated rotational ankle (AO/OTA 44 types A-C) fracture that is treated operatively
3. Abbreviated Injury Scale < 3 for non-extremity body systems
4. can speak, read, and understand English

Exclusion Criteria:

1. treated for a chronic pain condition prior to their qualifying injury
2. on a pain contract
3. pathologic fracture
4. Daily use of gabapentin or opiods prior to enrollment

Control Group:

Inclusion Criteria:

1. 18-85 years of age
2. can speak, read, and understand English

Exclusion Criteria:

1. Chronic pain or an ongoing acute pain condition
2. Currently or have previously sustained a bone fracture
3. Current Pain medication usage
4. Any previous orthopaedic surgical procedures
5. Must have been free of any surgeries for at least 5 years
6. Peripheral neuropathy
7. Individuals having had a major surgery or a major disease or condition, as determined by the PI, such as cardiovascular disease, metabolic disorders, renal disease, neurological disorders, or severe psychiatric conditions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will enroll participants who have sustained rotational ankle (specifically AO/OTA 44 types AC) fractures that are treated operatively. Fracture patients will complete clinic assessment sessions at standard of care visits, including their first post-op appointment (2-3 weeks), at 6-8 weeks, at 3-4 months, and at 6-9 months post-operatively. These visits will allow assessments during the subacute and chronic stages of bone fracture associated neuropathic pain.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Chronic Pain Grading Scale | 6-9 month
  Chronic Pain Grading Scale (CPGS) will be used to determine if fracture patients have pain in the chronic phase of injury (6-9 month visit). The pain intensity subscale will be used to categorize participants into those with and without chronic pain. This score is the sum of three questions (current pain, worst pain, average pain over last month), each scored on an 11-point Likert scale with responses ranging from 0-10 for a maximum of 30 points. The participant will be asked to report only on pain related to the site of fracture. Participants scoring 1-30 on the characteristic pain intensity score in the last month at the site of fracture will be classified as having chronic pain related to the fracture. Patients reporting no pain (0) at the site of fracture in the last month will be classified as having no chronic pain.
Douleur Neuropathique (Neuropathic Pain) 4 | 2 weeks to 1 year
  Douleur Neuropathique (Neuropathic Pain) 4 (DN4). The DN4 is a validated and reliable screening tool for neuropathic pain consisting of 10 items. The first 7 items relate to pain quality (i.e., sensory and pain descriptors) are based on interview with the patient. The last 3 items are based on clinical examination and assess hypoesthesia to touch, and hypoesthesia to prick and brushing. The items of the DN4 are scored based on a yes (1 point)/no (0 points) answer. This leads to a score range of 0-10. The cut-off value for the classification of neuropathic pain is a total score of 4 of 10.72 The DN4 has been used to identify NP in ankle fracture patients.
Assessment of Chronic Regional Pain Syndrome (CRPS) | 2 weeks to 6-9 months
  Assessment of Chronic Regional Pain Syndrome (CRPS). Presence of CRPS will be assessed in study participants beginning at the 6-8 week follow-up visit and all subsequent visits. Assessment of CRPS at earlier timepoints cannot be done rigorously as pain, motor, temperature and other changes comprising in part the CRPS diagnostic criteria can be related to the recent trauma. In addition to the QST procedures, a validated CRPS sign and symptom checklist will be administered by the study coordinator containing items in the 4 symptom and 4 sign categories needed to establish a CRPS diagnosis. For this study the investigators will employ the more rigorous CRPS Research Criteria (all symptom categories positive and 2/4 sign categories).
Central Sensitization measure | 5-9 weeks to 6-9 months
  Central Sensitization measure: The most common quantitative sensory test used to measure central sensitization in human experimental studies is temporal summation of pain (TS).TS will be administered on the skin proximal to the level of injury and the contralateral uninjured side using a nylon monofilament (Touchtest Sensory Evaluator 6.65) calibrated to bend at 300g of pressure. As in previous studies, participants will rate the perceived pain intensity of a single contact of the monofilament using a 0 to 100 numeric rating scale. Then, participants will provide another pain rating following a series of 10 contacts administered at a rate of 1 contact per second, applied to the body site within an area of 1 cm2. The difference between pain ratings for the single versus multiple contacts reflects temporal summation of mechanical pain. Two trials will be administered.
Pain Inhibitory Test | 5-9 weeks to 6-9 months
  Pain Inhibitory Test. Conditioned pain modulation (CPM) will be assessed by determining the ability of a cold pressor task to diminish pressure pain thresholds applied at a separate body site. For the conditioning stimulus, participants will immerse their non-affected hand up to the wrist in a cold water bath maintained at 10 degrees C for up to 1 minute or until they report intolerable pain.The test stimulus will be two trials of pressure pain thresholds (PPTs) administered on the left forearm. The experimenter will apply a slow constant rate of pressure and the participant will press a button when the sensation first becomes painful, at which time a device records the pressure. Three consecutive measurements with intervals of 20s will be obtained pre- and post- the conditioning stimulus.

SECONDARY OUTCOMES:
Mechanical Detection Thresholds | 5-9 weeks to 6-9 months
  Mechanical detection thresholds will be examined using von Frey monofilaments, with each filament applied three times in ascending sequence until the threshold is detected in at least two of the three trials. Then, the next lower von Frey filament will be applied, and the lowest filament to be detected at least twice will be determined as the mechanical detection threshold.
Pressure pain thresholds | 5-9 weeks to 6-9 months
  A digital, handheld, clinical grade pressure algometer will be used for the mechanical procedures (AlgoMed, Medoc). The experimenter will apply a slow constant rate of pressure and record the pressure in kilograms when the subject responds. Pressure will be applied using a .5 cm2 probe. Subjects will be instructed to respond when they first feel pain and pressure at threshold will be recorded. Two consecutive measurements at each point with intervals of 20 s will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Roman Natoli, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Johansen A, Romundstad L, Nielsen CS, Schirmer H, Stubhaug A. Persistent postsurgical pain in a general population: prevalence and predictors in the Tromso study. Pain. 2012 Jul;153(7):1390-1396. doi: 10.1016/j.pain.2012.02.018. Epub 2012 Mar 24. PMID 22445291
- [Background] Scheer RC, Newman JM, Zhou JJ, Oommen AJ, Naziri Q, Shah NV, Pascal SC, Penny GS, McKean JM, Tsai J, Uribe JA. Ankle Fracture Epidemiology in the United States: Patient-Related Trends and Mechanisms of Injury. J Foot Ankle Surg. 2020 May-Jun;59(3):479-483. doi: 10.1053/j.jfas.2019.09.016. PMID 32354504
- [Background] Karl JW, Olson PR, Rosenwasser MP. The Epidemiology of Upper Extremity Fractures in the United States, 2009. J Orthop Trauma. 2015 Aug;29(8):e242-4. doi: 10.1097/BOT.0000000000000312. PMID 25714441
- [Background] Beetar JT, Guilmette TJ, Sparadeo FR. Sleep and pain complaints in symptomatic traumatic brain injury and neurologic populations. Arch Phys Med Rehabil. 1996 Dec;77(12):1298-302. doi: 10.1016/s0003-9993(96)90196-3. PMID 8976315
- [Background] Veljkovic A, Dwyer T, Lau JT, Abbas KZ, Salat P, Brull R. Neurological Complications Related to Elective Orthopedic Surgery: Part 3: Common Foot and Ankle Procedures. Reg Anesth Pain Med. 2015 Sep-Oct;40(5):455-66. doi: 10.1097/AAP.0000000000000199. PMID 26192548
- [Background] Rbia N, van der Vlies CH, Cleffken BI, Selles RW, Hovius SER, Nijhuis THJ. High Prevalence of Chronic Pain With Neuropathic Characteristics After Open Reduction and Internal Fixation of Ankle Fractures. Foot Ankle Int. 2017 Sep;38(9):987-996. doi: 10.1177/1071100717712432. Epub 2017 Jul 1. PMID 28670914
- [Background] Nahin RL. Severe Pain in Veterans: The Effect of Age and Sex, and Comparisons With the General Population. J Pain. 2017 Mar;18(3):247-254. doi: 10.1016/j.jpain.2016.10.021. Epub 2016 Nov 21. PMID 27884688
- [Background] Vallerand AH, Cosler P, Henningfield JE, Galassini P. Pain management strategies and lessons from the military: A narrative review. Pain Res Manag. 2015 Sep-Oct;20(5):261-8. doi: 10.1155/2015/196025. PMID 26448972
- [Background] Baca Q, Marti F, Poblete B, Gaudilliere B, Aghaeepour N, Angst MS. Predicting Acute Pain After Surgery: A Multivariate Analysis. Ann Surg. 2021 Feb 1;273(2):289-298. doi: 10.1097/SLA.0000000000003400. PMID 31188202
- [Background] Sun S, Diggins NH, Gunderson ZJ, Fehrenbacher JC, White FA, Kacena MA. No pain, no gain? The effects of pain-promoting neuropeptides and neurotrophins on fracture healing. Bone. 2020 Feb;131:115109. doi: 10.1016/j.bone.2019.115109. Epub 2019 Nov 9. PMID 31715336
- [Background] Lamparello AJ, Namas RA, Constantine G, McKinley TO, Elster E, Vodovotz Y, Billiar TR. A conceptual time window-based model for the early stratification of trauma patients. J Intern Med. 2019 Jul;286(1):2-15. doi: 10.1111/joim.12874. Epub 2019 Jan 9. PMID 30623510
- [Background] McKinley TO, Gaski GE, Zamora R, Shen L, Sun Q, Namas RA, Billiar TR, Vodovotz Y. Early dynamic orchestration of immunologic mediators identifies multiply injured patients who are tolerant or sensitive to hemorrhage. J Trauma Acute Care Surg. 2021 Mar 1;90(3):441-450. doi: 10.1097/TA.0000000000002998. PMID 33093290
- [Background] Almahmoud K, Abboud A, Namas RA, Zamora R, Sperry J, Peitzman AB, Truitt MS, Gaski GE, McKinley TO, Billiar TR, Vodovotz Y. Computational evidence for an early, amplified systemic inflammation program in polytrauma patients with severe extremity injuries. PLoS One. 2019 Jun 4;14(6):e0217577. doi: 10.1371/journal.pone.0217577. eCollection 2019. PMID 31163056